CLINICAL TRIAL: NCT00635934
Title: A Prospective, Non-Randomized Pilot Clinical Investigation of the A-MAV™ Anterior Motion Segment Replacement in Patients With Lumbar Degenerative Disc Disease
Brief Title: A-MAV™ Anterior Motion Segment Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04-05
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2011-10

CONDITIONS: Spinal Diseases
Keywords: Lumbar Degenerative Disc Disease at One Level from L4-S1
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A-MAV™disc (Experimental)
  Interventions: Device: A-MAV™ disc

INTERVENTIONS:
Device: A-MAV™ disc — The A-MAV™ device is a spinal arthroplasy system intended to replace a damaged spinal disc. It is inserted using an anterior surgical approach and aims to reduce low back pain and maintain disc height at the affected level.
  Other Names: A-MAV™

SUMMARY:
The purpose of this clinical trial is to collect safety and effectiveness data concerning the A-MAV™ Anterior Motion Segment Replacement device as a method of treating patients with lumbar degenerative disc disease at one level from L4-S1. Overall success will be the primary clinical endpoint.

DETAILED DESCRIPTION:
For this clinical trial, there is only one treatment group- patients receiving the A-MAV™ Anterior Motion Segment Replacement via an anterior surgical approach in the lumbar region of the spine from L4-S1.

ELIGIBILITY:
Inclusion Criteria:

* Has back and/or radicular pain with degeneration of the disc as confirmed by patient history, physical examination, and radiographic studies with one or more of the following factors:

  * instability as defined by > 5° angulation
  * osteophyte formation of facet joints or vertebral endplates
  * decreased disc height, on average by >2mm, relative to the next adjacent vertebral segment
  * scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule
  * herniated nucleus pulposus
  * facet joint degeneration/changes
  * vacuum phenomenon
* Has single-level symptomatic degenerative involvement from L4-S1 requiring surgical treatment
* Has intact facet joints at the involved vertebral levels documented by CT and/or MRI
* Has preop Oswestry score≥30
* Has preop back pain score ≥8
* Age 18 to 70 yrs, inclusive and is skeletally mature
* Has not responded to non-operative treatment for 6 mos
* If child-bearing potential, patient is non-pregnant, non-nursing, and agrees not to become pregnant for 1 yr after surgery
* Is willing and able to comply with the study plan and sign the Patient Informed Consent Form

Exclusion Criteria:

* Has primary diagnosis of a spinal disorder other than DDD at involved level
* Had previous anterior lumbar spinal surgery at involved level
* Had previous posterior lumbar spinal fusion surgical procedure at involved level
* Had prior posterior lumbar surgery resulting in significant muscle/ligament morbidity, not including facet saving techniques
* Requires surgical intervention at more than 1 lumbar level
* Has severe pathology of facet joints of involved vertebral bodies
* Has facet arthritis or any posterior element insufficiency
* Has spondylolisthesis
* Has mid-sagittal stenosis of <8mm, based on remaining canal diameter
* Has rotatory scoliosis at involved level
* Has lumbar scoliosis with >11° sagittal plane deformity
* Had previous trauma to L4, L5, or S1 levels in compression or burst
* Meets any of the following criteria: Previous diagnosis of osteoporosis, osteopenia, or osteomalacia; postmenopausal Non-Black female over 60 yrs of age and weighs less than 140 pounds; postmenopausal female that has sustained a non-traumatic hip, spine or wrist fracture; male over age 60 that has sustained a non-traumatic hip or spine fracture. If Yes to any of these, a DEXA scan is required. If level of BMD is -3.5 or lower or -2.5 or lower with vertebral crush fracture, the patient is excluded
* Had previous lumbar spinal fusion at adjacent level
* Bone growth stimulator use in spine
* Has obesity defined by BMI greater than or equal to 40
* Has arachnoiditis
* Has a non-contained or extruded herniated nucleus pulposus with acute nerve root compression
* Has condition that requires postop medications that interfere with bone metabolism, such as chronic steroid use or prolonged use of non-steroidal anti-inflammatory drugs, excluding routine perioperative, non-steroidal anti-inflammatory drugs. Does not include low dose aspirin for prophylactic anticoagulation
* Has overt or active bacterial infection, either local or systemic and/or potential for bacteremia
* Has presence or prior history of malignancy (except for basal cell carcinoma of skin)
* Has documented metal allergy, titanium alloy intolerance or cobalt-chrome-molybdenum alloy
* Is mentally incompetent. If questionable, obtain psych consult
* Has a Waddell Signs of Inorganic Behavior score of 3 or greater
* Has chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease
* Is prisoner
* Is pregnant
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse
* Has history of autoimmune disease
* Has received treatment with an investigational therapy within 30 days prior to implantation surgery or treatment is planned during 24 months following the implantation surgery
* Has history of any endocrine or metabolic disorder known to affect osteogenesis
* Has any disease that would preclude accurate clinical evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Overall Success= Oswestry Disability Index success; Maintenance or improvement in neurological status; No serious AE classified as implant or implant/surgical procedure associated; No additional surgical procedure classified as a failure | 24 Months

SECONDARY OUTCOMES:
Disc height; SF-36; Back Pain Status; Leg Pain Status; Patient Satisfaction; Patient Global Perceived Effect; Other Measurements-Radiographic; Return to Work; Doctor's Perception of Results | 24 Months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hughston Clinic, Columbus, Georgia
  - Orthopedic Center of St. Louis, Chesterfield, Missouri
  - Central Texas Spine, Austin, Texas